CLINICAL TRIAL: NCT01883232
Title: The Efficacy of Analgesic Buffering With Sodium Bicarbonate for the Pediatric Dental Patient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0298
Record Dates: First submitted 2013-05-17; First posted 2013-06-21 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2% lidocaine with 1:100,000 epinephrine (Active Comparator): 2% lidocaine with 1:100,000 epinephrine
  Interventions: Device: 2% lidocaine with 1:100,000 epinephrine
- Onset Mixing Pen by Onpharma (Experimental): Sodium Bicarbonate 8.4% mixed with the onset mixing pen
  Interventions: Device: Onset Mixing Pen by Onpharma

INTERVENTIONS:
Device: Onset Mixing Pen by Onpharma — Sodium Bicarbonate 8.4%
  Arms: Onset Mixing Pen by Onpharma
Device: 2% lidocaine with 1:100,000 epinephrine — 2% lidocaine with 1:100,000 epinephrine administered with a syringe prior to the procedure
  Arms: 2% lidocaine with 1:100,000 epinephrine

SUMMARY:
As a dentist, administering anesthetic to patients, especially children, proves to be one of the most difficult parts of a procedure. Pain is one of the most common symptom in dentistry, and a serious concern for the dentist. The pain of the local anesthetic injection has several causes. Of the many reasons for pain at the site of injection, the acidity of the solution is thought to be most important. This study will be measuring the effects of adding sodium bicarbonate (buffer) to local anesthetic during dental procedures. This is commonly used in medical applications but is not widely used in the dental setting. Using this biochemistry and human physiology, one can predict when buffering the lidocaine injection, a quicker response in analgesia and a decrease in pain during administration. I will be measuring the effect using several measuring devices to gauge if buffering the local anesthetic will benefit the pediatric dental patient by reducing the time it takes for the analgesic effect as well as decreasing the pain during administration. Along with time, I will be using the Wong-Baker Scale to assess the pain. This scale is standard protocol for assessing pain in the pediatric population. The pediatric dental population has aversions to dental procedures because of the associated pain produced from most procedures. If limiting the time it takes for the analgesic to take effect and decrease the pain altogether, the pediatric patient will be less likely to skip treatment therefore, increase dental health.

ELIGIBILITY:
Inclusion Criteria:

* Current patients of Children's Hospital Colorado Dental Clinic
* Existence of carious primary molars necessitating administration of an anesthetic agent
* No history of post traumatic stress disorder or specific phobia related to a dental setting
* No allergic reaction to lidocaine
* Patient's between the ages of 5 to 12.

Exclusion Criteria:

* Allergies to local anesthetics or sulfites
* History of significant medical conditions
* Taking any medications that may affect anesthetic assessment
* Active sites of pathology in areas if injection
* Outside the age range of 5 -12.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in pain rating using the Wong-Baker scale | During injection (about 5 minutes)
  By buffering the lidocaine/epinephrine injection, one should see a decrease in in pain during the administration of the anesthetic.
Time it takes for buffered injection to take effect measured in minutes. | 5 minutes
  minutes for the analgesic effect to take place.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Esker, DMD, Principal Investigator — Children's Hospital Colorado Dental Clinic
Locations (1):
- Children's Hospital Colorado Dental Clinic, Aurora, Colorado, United States

REFERENCES:
- [Result] Kashyap VM, Desai R, Reddy PB, Menon S. Effect of alkalinisation of lignocaine for intraoral nerve block on pain during injection, and speed of onset of anaesthesia. Br J Oral Maxillofac Surg. 2011 Dec;49(8):e72-5. doi: 10.1016/j.bjoms.2011.04.068. Epub 2011 May 18. PMID 21592633
- [Result] Grassick P. The fear behind the fear: a case study of apparent simple injection phobia. J Behav Ther Exp Psychiatry. 1990 Dec;21(4):281-7. doi: 10.1016/0005-7916(90)90030-o. PMID 1982735
- [Result] Arndt KA, Burton C, Noe JM. Minimizing the pain of local anesthesia. Plast Reconstr Surg. 1983 Nov;72(5):676-9. doi: 10.1097/00006534-198311000-00017. PMID 6622575
- [Result] Meit SS, Yasek V, Shannon CK, Hickman D, Williams D. Techniques for reducing anesthetic injection pain: an interdisciplinary survey of knowledge and application. J Am Dent Assoc. 2004 Sep;135(9):1243-50. doi: 10.14219/jada.archive.2004.0399. PMID 15493388
- [Result] Burns CA, Ferris G, Feng C, Cooper JZ, Brown MD. Decreasing the pain of local anesthesia: a prospective, double-blind comparison of buffered, premixed 1% lidocaine with epinephrine versus 1% lidocaine freshly mixed with epinephrine. J Am Acad Dermatol. 2006 Jan;54(1):128-31. doi: 10.1016/j.jaad.2005.06.043. PMID 16384767
- [Result] Reed KL, Malamed SF, Fonner AM. Local anesthesia part 2: technical considerations. Anesth Prog. 2012 Fall;59(3):127-36; quiz 137. doi: 10.2344/0003-3006-59.3.127. PMID 23050753
- [Result] Malamed SF, Falkel M. Advances in local anesthetics: pH buffering and dissolved CO2. Dent Today. 2012 May;31(5):88-93; quiz 94-5. No abstract available. PMID 22650087
- [Result] Christoph RA, Buchanan L, Begalla K, Schwartz S. Pain reduction in local anesthetic administration through pH buffering. Ann Emerg Med. 1988 Feb;17(2):117-20. doi: 10.1016/s0196-0644(88)80293-2. PMID 2827545
- [Result] Aminabadi NA, Farahani RM, Balayi Gajan E. The efficacy of distraction and counterstimulation in the reduction of pain reaction to intraoral injection by pediatric patients. J Contemp Dent Pract. 2008 Sep 1;9(6):33-40. PMID 18784857